CLINICAL TRIAL: NCT06689306
Title: TEACHING CARE BEHAVIORS to NURSING STUDENTS WITHIN the 7E LEARNING MODEL: a RANDOMIZED CONTROLLED STUDY
Brief Title: 7E Model in Nursing Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sema Köse, Ataturk Universty, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: sema_kose_doktora_tezi
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Nursing Education; Nursing Care
Keywords: Nursing; nursing care; nursing education; human caring theory; 7E model

STUDY DESIGN:
Intervention Model Description: The sample of the study consists of 70 second-year nursing students studying at the Nursing Department of the Faculty of Health Sciences at Erzincan Binali Yıldırım University, who have chosen the Development of Caring Behaviors course as an elective course and will be divided into sections A and B (without any intervention) through the system. In the study, one section will be selected by flipping a coin by someone other than the researcher using the simple randomization method and the other section will be the experimental group and the other section will be the control group. The study will be designed so that the students will not know whether they are in the intervention or control group, and one-way blinding will be applied in the study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Necessary explanations regarding the research will be made to the students and their verbal and written consents will be obtained.
  * Application Week 1: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) Pre-Test Applications
  * In the 2nd, 3rd, 4th and 5th weeks, the topic of developing care behaviors will be covered with the 7E model.
  * Application Week 7: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) post-test applications
  * Application Week 11: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) follow-up test applications
  Interventions: Behavioral: 7E learning model
- Control group (No Intervention): The necessary explanations about the research will be made to the students and their verbal and written consents will be obtained.
  * Application Week 1: "Descriptive Information Form (DEF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) Pre-Test Applications
  * The topic of developing care behaviors in the 2nd, 3rd, 4th and 5th weeks will be handled through plain narration and question-answer methods.
  * Application Week 7: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) post-test applications
  * Application Week 11: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) follow-up test applications

INTERVENTIONS:
Behavioral: 7E learning model — 7E learning model7E learning cycle is a teaching model that encourages students to be active, to think about the findings they obtain, to interpret their findings according to their initial plans and to predict them in new situations. This model provides students with opportunities for discussion and interaction. The model is designed based on constructivist theory. The guiding concept of constructivism is that later learning is greatly influenced by previous knowledge; therefore, learning should be based on the interaction of old and new knowledge. 7E learning cycle model consists of seven steps: Reveal, Participate, Explore, Explain, Elaborate, Evaluate and Extend. According to past studies, 7E model is more effective in developing students than traditional learning models.
  Arms: Experimental group

SUMMARY:
This study aimed to examine the effects of teaching caring behaviors based on the 7E learning model on nursing students' course success, learning permanence, critical thinking skills and motivation levels.

DETAILED DESCRIPTION:
This research is a randomized controlled experimental study aiming to evaluate the effect of the intervention. The research data were planned to be collected from second-year nursing students studying at the Nursing Department of the Faculty of Health Sciences at Erzincan Binali Yıldırım University between October 2024 and January 2025. The Development of Caring Behaviors Course will be conducted by the researcher in two different sections in this faculty in the fall semester. The student quota for each section was determined as 35. The universe of the research will consist of second-year students studying in the nursing department of a state university. There are a total of 136 students in the second year of nursing. Second-year nursing students who selected the Development of Caring Behaviors Course as an elective course and agreed to participate in the research (two different sections, 70 students) will constitute the sample of the research. In the study, one branch selected by simple random method will constitute the experimental group and one branch will constitute the control group.

The sample of the study consists of 70 second-year nursing students studying at Erzincan Binali Yıldırım University, Faculty of Health Sciences, Department of Nursing, who have chosen the Development of Caring Behaviors course as an elective course and will be divided into sections A and B through the system (without any intervention). In the study, one branch selected by flipping a coin by someone other than the researcher with simple randomization method will constitute the experimental group and one branch will constitute the control group. The study will be designed in a way that students will not know whether they are in the intervention or control group, and one-way blinding will be applied in the study. The data of the study will be collected using the "Diagnostic Information Form (DIF)" including the socio-demographic characteristics of the individuals created in line with the literature, the "Academic Achievement Test (ABT)" prepared specifically for the subjects to evaluate course success and permanence of learning, the California Critical Thinking Disposition Scale (CCTDS), and the Instructional Materials Motivation Survey (IMMS) The research will be conducted in Erzincan between October 2024 and January 2025. It will be conducted in the Development of Caring Behaviors course of second-year nursing students of a state university. The researcher (SK) works as a lecturer at this school. The development of caring behaviors course is an elective course opened in the fall semester for second-year nursing students and the class quota of the course is determined as 35. The researcher (SK) conducts this course alone.

In the content plan of the Development of Caring Behaviors Course, the topics of caring behaviors are given in five weeks. The topics given in the following weeks differ. Therefore, the implementation plan of the research was made for the first weeks of the course.

In the research, one branch selected by flipping a coin by someone other than the researcher with the simple randomization method will constitute the experimental group and one branch will constitute the control group. The research will be designed in a way that the students will not know whether they are in the intervention or control group, and one-way blinding will be applied in the research.

Control Group:

The necessary explanations about the research will be made to the students and their verbal and written consents will be obtained.

* Application Week 1: "Descriptive Information Form (DEF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) Pre-Test Applications
* Application Week 2: The Concept of Care and Human Care Theory and Care Behaviors topics will be covered with plain narration and question-answer methods.
* Application Week 3: Care Behaviors: Care Situation and Care Moment, Interpersonal Care Relationship topics will be covered with plain narration and question-answer methods.
* Application Week 4: Care Behaviors: Being Present, Presenting Your Presence topics will be covered with plain narration and question-answer methods.
* Application Week 5: Care Behaviors: Being Present, Presenting Your Presence, Authentic Listening topics will be covered with plain narration and question-answer methods.
* Application Week 6: Care Behaviors: Accepting the Individual, Making Eye Contact, Addressing by Name, Smiling, Touching will be covered with plain narration and question-answer methods.
* Application Week 7: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) post-test applications
* Application Week 11: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) follow-up test applications

Experimental Group:

Necessary explanations regarding the research will be made to the students and their verbal and written consents will be obtained.

* Application Week 1: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) Pre-Test Applications
* Application Week 2: The Concept of Care and Human Care Theory and Care Behaviors will be covered with the 7E model.
* Application Week 3: Care Behaviors: Care Situation and Care Moment, Interpersonal Care Relationship topics will be covered with the 7E model.
* Application Week 4: Care Behaviors: Being Present, Offering Your Presence topics will be covered with the 7E model.
* Application Week 5: Care Behaviors: Being Present, Offering Your Presence, Authentic Listening topics will be covered with the 7E model.
* Application Week 6: Care Behaviors: Accepting the Individual, Making Eye Contact, Addressing by Name, Smiling, Touching topics will be covered with the 7E model.
* Application Week 7: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) post-test applications
* Application Week 11: "Diagnostic Information Form (DIF)", "Academic Achievement Test" (ABT), California Critical Thinking Disposition Scale (CCTDS), Instructional Materials Motivation Survey (IMMS) follow-up test applications 7E learning cycle model consists of seven steps: Engage, eliciting, explore, explain, elaborate, evaluate, and relate. Maintenance behaviors Subject contents will be prepared by addressing these seven steps. Active learning methods (talking circle, thought walk, 6 (Six) Thinking Hats Method, concept map, etc.) suitable for each step and subject content will be used in the implementation of the course.

To evaluate the effect of the training intervention, all participants will fill out all data collection forms for the third time for the follow-up test one month after the training intervention. A one-month break is planned for the follow-up test in order to avoid the test effect.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Not having dealt with this topic before,
* Being a second year nursing student
* Being willing to participate in the study
* Not having any communication barriers,
* Not having a psychiatric illness diagnosis or treatment.

Exclusion Criteria:

* The student is from upper grades and taking this course from lower grades
* Being a foreign national
* Not wanting to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
H1- Using the 7E learning model in teaching caring behaviors affects the course success of nursing students. | one week before, one week after completion
  An academic achievement test will be administered to participating students one week before starting the care behaviors education in line with the 7E learning model and one week after the training is completed.
H2- Using the 7E learning model in teaching caring behaviors affects the permanent learning of nursing students. | 5 weeks after completion of training
  An academic achievement test will be administered to participating students one week before starting the care behaviors training in line with the 7E learning model and 5 weeks after the training is completed.
H3- The use of the 7E learning model in teaching caring behaviors affects the motivation levels of nursing students. | one week before, one week after completion of training and 5 weeks after completion of training
  Instructional Materials Motivation Survey (IMMS) will be administered to the participating students three times: one week before starting the care behaviors teaching given in line with the 7E learning model, one week after the training was completed, and five weeks after the training was completed.
H4- The use of the 7E learning model in teaching caring behaviors affects the critical thinking skills of nursing students. | one week before, one week after completion of training and 5 weeks after completion of training
  The California Critical Thinking Disposition Scale (CCTDS) will be administered to participating students three times: one week before starting the care behaviors education given in line with the 7E learning model, one week after the completion of the training, and 5 weeks after the completion of the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Başbağlar neighborhood 1410 street Faculty of Health Sciences Center Erzincan, Erzincan Merkez, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No